CLINICAL TRIAL: NCT06867081
Title: Effectiveness of a Customized Digital Platform to Increase Coordination of Care and Uptake of Evidence-based Practices: a Protocol for a Stepped-wedge Cluster Randomized Trial in Quebec
Brief Title: Effectiveness of a Customized Digital Platform to Increase Coordination of Care and Uptake of Evidence-based Practices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Sara Ahmed, Principal Investigator, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-58314; 481022 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-11-01; First posted 2025-03-10 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Aquired Brain Injury; Traumatic Brain Injuries; Stroke; Cardiovascular Diseases
Keywords: Acquired brain injury; Digital health platform; Rehabilitation; Transition of care; Person-centered care; Implementation science; stepped wedge trial
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Cardiovascular Diseases; Brain Injuries

STUDY DESIGN:
Intervention Model Description: We will conduct a stepped wedge cluster randomized trial in four health regions and 8 programs (i.e., clusters).
  A stepped wedge cluster randomized trial is a special case of cluster cross over designs particularly useful in an educational context where clusters (e.g., programs, clinicians) can only change their exposure status (i.e., participation in the intervention) in one direction (i.e., from less knowledgeable, before the intervention, to more knowledgeable, after the intervention). It is an ideal design as programs intend to implement the BRILLIANT platform as an ongoing part of practice. We expect trends over time will be similar across all ABI programs in each region. Identification and recruitment bias is a concern in stepped wedge trials when recruitment occurs after randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Rehabilitation Program 1 (Experimental): The program provides intensive rehabilitation following ABI guidelines and in line with other provinces and countries. There is a period when outcomes are collected during an initial control period (2 to 7 months depending on when the program is randomized to receive the intervention), followed by an intervention period when the digital health platform is deployed (12 months to 22 months depending on when the program is randomized).
  Interventions: Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time
- Rehabilitation Program 2 (Experimental): The program provides intensive rehabilitation following ABI guidelines and in line with other provinces and countries. There is a period when outcomes are collected during an initial control period (2 to 7 months depending on when the program is randomized to receive the intervention), followed by an intervention period when the digital health platform is deployed (12 months to 22 months depending on when the program is randomized).
  Interventions: Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time
- Rehabilitation Program 3 (Experimental): The program provides intensive rehabilitation following ABI guidelines and in line with other provinces and countries. There is a period when outcomes are collected during an initial control period (2 to 7 months depending on when the program is randomized to receive the intervention), followed by an intervention period when the digital health platform is deployed (12 months to 22 months depending on when the program is randomized).
  Interventions: Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time
- Rehabilitation Program 4 (Experimental): The program provides intensive rehabilitation following ABI guidelines and in line with other provinces and countries. There is a period when outcomes are collected during an initial control period (2 to 7 months depending on when the program is randomized to receive the intervention), followed by an intervention period when the digital health platform is deployed (12 months to 22 months depending on when the program is randomized).
  Interventions: Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time
- Rehabilitation Program 5 (Experimental): The program provides intensive rehabilitation following ABI guidelines and in line with other provinces and countries. There is a period when outcomes are collected during an initial control period (2 to 7 months depending on when the program is randomized to receive the intervention), followed by an intervention period when the digital health platform is deployed (12 months to 22 months depending on when the program is randomized).
  Interventions: Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time
- Rehabilitation Program 6 (Experimental): The program provides intensive rehabilitation following ABI guidelines and in line with other provinces and countries. There is a period when outcomes are collected during an initial control period (2 to 7 months depending on when the program is randomized to receive the intervention), followed by an intervention period when the digital health platform is deployed (12 months to 22 months depending on when the program is randomized).
  Interventions: Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time
- Rehabilitation Program 7 (Experimental): The program provides intensive rehabilitation following ABI guidelines and in line with other provinces and countries. There is a period when outcomes are collected during an initial control period (2 to 7 months depending on when the program is randomized to receive the intervention), followed by an intervention period when the digital health platform is deployed (12 months to 22 months depending on when the program is randomized).
  Interventions: Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time
- Rehabilitation Program 8 (Experimental): The program provides intensive rehabilitation following ABI guidelines and in line with other provinces and countries. There is a period when outcomes are collected during an initial control period (2 to 7 months depending on when the program is randomized to receive the intervention), followed by an intervention period when the digital health platform is deployed (12 months to 22 months depending on when the program is randomized).
  Interventions: Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time

INTERVENTIONS:
Other: The intervention will be the BRILLIANT Platform, an online platform which provides five Modules aimed at increasing coordination of care and direct rehabilitation time — The BRILLIANT Platform provides five Modules aimed at increasing coordination of care and direct rehabilitation time: 1) Standardized measures: provided consistently with scoring and reminders to complete assessments, across all stages of recovery and care settings to guide and evaluate treatment effectiveness of clinical outcomes, performance based outcomes, patient reported outcome measures; 2) Communication Module: clinicians can communicate together and with patient/family to clarify patient-related information and update colleagues for time sensitive information, synchronously and asynchronously; 3) Shared intervention goals and plan: personalized and dynamic care trajectory and intervention plan guided by standardized assessments, reminders, and evidence-based interventions recommendations to direct patients and caregivers to the right services and interventions at the right time based on clinical and social profile and best practices; and 2 other related topics.

SUMMARY:
Background: Cardiovascular and neurological conditions are major causes of disability worldwide. Early, intensive rehabilitation is essential but often challenging to access in current healthcare systems. In Canada, the direct and indirect costs of acquired brain injury (ABI) are substantial, emphasizing the need for improved rehabilitation services. In collaboration with four health regions and the Canadian Foundation of Innovation (CFI) funded BRILLIANT research group, investigators are implementing a digital health platform (the BRILLIANT platform), which includes five modules to address current gaps and support a person-centered integrated care continuum for cardiovascular and neurological conditions. In this stepped wedge randomized trial, investigators plan to implement and evaluate the use of the BRILLIANT Platform for improving transitions of care in the rehabilitation of ABI individuals in Quebec.

Methods: A stepped wedge cluster randomized trial will be conducted across four healthcare regions with eight programs. Eligible participants included new cardiovascular and neurological patients, caregivers, clinicians, coordinators, and managers. The BRILLIANT platform intervention, implemented in 2 phases, will provide standardized assessments, communication tools, shared intervention plans, self-management support, and quality improvement dashboards. Outcomes will include rehabilitation intensity measured in minutes, time from admission to rehabilitation, health-related quality of life, care experience, and costs. Data analysis will use mixed-effects models for quantitative data and content analysis for qualitative data.

Discussion: This study will provide valuable evidence on the effectiveness and feasibility of the BRILLIANT platform in improving rehabilitation care for patients with cardiovascular and neurological conditions in Quebec. Investigators anticipate that by addressing the challenges and pursuing future directions, the implementation of this digital platform can contribute to improving patient outcomes and healthcare delivery.

DETAILED DESCRIPTION:
Research questions and sites The research questions guiding this study are: 1) What are the potential barriers and facilitators in the implementation of the BRILLIANT platform at the local teams' level?; 2) What is the impact of the BRILLIANT platform compared to usual cardiovascular and neurological care on the primary outcome, intensity of rehabilitation (direct minutes of rehabilitation per week); 3) Does the platform have an impact on secondary outcomes: time to be admitted to rehabilitation (inpatient or outpatient), health-related quality of life, care experience, and if found to be effective, costs?; 4) What are the implementation factors that explain potential impact (e.g., relevance, acceptability)? An integrated knowledge translation (iKT) approach will be used by involving all relevant partners throughout the research process. The partners are stakeholders within four health regions with two to four programs each in various rehabilitation stages for cardiovascular and neurological care in Quebec. In four health regions and 8 cardiovascular and neurological programs, this implementation study follows two phases aiming answering the 4 research questions.

Study phases and procedures Phase I is for measuring and addressing the potential barriers and facilitators related to the implementation of the BRILLIANT platform and prepare teams for implementation. With each program investigators will review the workflow (clinical processes and the material and human resources available) for cardiovascular and neurological care pathways, and use the Business Process Model and Notation (BPMN) method and analyze them to maximize successful implementation during the trial. The purpose of this first phase is to determine what the BRILLIANT platform will look like. Through focus groups with 8-10 participants per program comprised of all health professions, coordinators, managers, and patient/family participants with experience with different phases of the rehabilitation process. In the focus groups, investigators will review how the platform will work, validate certain tasks, and ensure ease of use so that investigators may adjust as needed. Identifying barriers and facilitators to implementing the platform during the focus groups will be guided by the Consolidated Framework for Implementation Research (CFIR). Focus group sessions will be recorded and transcribed, and further analysed to feed back information on barriers and facilitators during subsequent design workshops to also inform adaptation and implementation of the platform.

The second phase is to evaluate the impact of the BRILLIANT platform on primary (intensity of rehabilitation, i.e. direct minutes of rehabilitation per week), and secondary outcomes (time to be admitted to inpatient or outpatient rehabilitation, health-related quality of life, care experience, and costs if the platform is found to have an impact) and evaluating the factors that impact implementation. The control condition will be usual care, which consists of an interdisciplinary team of physiotherapy, occupational therapy, nursing, medicine, psychology, speech therapy, social work, and nutrition. Clinicians mostly work on paper evaluating patient needs (mostly by checklist) using static standardized forms (e.g., Functional Independence Measure, FIM, at admission) without reminders, scoring and interactive functionalities. The choice of standardized assessment is left to the discretion of each clinician. Since the pandemic Microsoft teams is used to share scanned documents between clinicians and remote program meetings. During the control period clinicians will have access to static forms on the BRILLIANT Platform.

Intervention details The intervention will be the use of the BRILLIANT Platform. The platform provides five Modules aimed at increasing coordination of care and direct rehabilitation time (Table 1): 1) Standardized measures: provided consistently with scoring and reminders to complete assessments, across all stages of recovery and care settings to guide and evaluate treatment effectiveness of clinical outcomes (e.g. FIM, Mayo Portland Adaptability Inventory - MPAI), performance based outcomes (e.g. gait speed), patient reported outcome measures (e.g. pain level during walking); 2) Communication Module: clinicians can communicate together and with patient/family to clarify patient-related information (e.g. safety concerns, intervention plan progression) and update colleagues for time sensitive information, synchronously (scheduled tele-videoconference) and asynchronously; 3) Shared intervention goals and plan: personalized and dynamic care trajectory and intervention plan guided by standardized assessments, reminders, and evidence-based interventions recommendations to direct patients and caregivers to the right services and interventions (e.g. treadmill walking practice) at the right time based on clinical and social profile and best practices;1,2 4) Self-management support: To provide patients and families with self-management dashboards (e.g. physical activity tracking and reminders) and interactive online intervention plan (goals, action plan, monitoring progress) to actively engage the patient and family in setting goals with their care team. Access to evidence-based patient education and resource modules, tailored to stage of recovery (e.g. Education on how to handle arm or shoulder); 5) Quality Improvement Dashboards to provide feedback and reports allowing observation of clinical/administrative/clinical performance indicators (based on MSSS indicators, Quadruple Aim framework) for continuous program evaluation.

Each health region will be provided with cloud-based access to the platform as agreed in collaboration with their IT units. Each site will have support from a knowledge broker from the research team to promote the platform's purpose, features and benefits and build understanding, and engagement of the local programs. Pre-implementation, there will be: 1) a 2-hour training session (respecting COVID restrictions) in each site and an online training video that participants can access anytime; 2) a platform guidebook explaining each functionality, that can be accessed anytime.

Based on ongoing implementation of new practices in these programs the investigators will use the following six evidence-based implementation strategies: 1) organize implementation meetings; 2) provide educational materials (e.g. videos) on platform use; 3) conduct ongoing training for new platform users; 4) audit and feedback of optimal use indicators to platform users; 5) engage health region digital health leads in the implementation process; 6) provide local assistance for rapid resolution of technical issues. The duration of follow up is 12 months to allow time for sites to practice and adopt the platform and increase likely impact on change in rehabilitation intensity and outcomes given the recovery and clinical process post ABI. Twelve months are necessary to account for differences across sites that stem from admission rates.

Randomization After a period of 2 months, when all programs have access to the BRILLIANT platform only with static forms (control), randomisation of the first 2 sites will start. Programs will enter the trial in four consecutive waves based on stratified randomisation controlling for health region and type of program (cardiovascular or neurological). This will help to minimise, in part, temporal trends due to region and program, if any exist. Each step will enroll 2 programs at a time (paired stepped-wedge), to allow the training and trouble-shooting period to take place in a limited number of sites at a time. The enrolment process will take 27 months, allowing for a minimum 12-month follow-up in the last two programs receiving the intervention. Programs will receive sufficient notice of the dates to cross over to the intervention.

Knowledge Translation Plan The four health regions, patient, and industry partners have outlined their commitment to this project. The investigators will have knowledge exchange sessions between health regions to share best practices throughout all phases of the project. The iKT and Living lab approach entails continuous co-creation and exchange throughout the study. For this study, the primary end-of-grant KT activities will consist of 1) a stakeholder-generated report integrating all our findings; and 2) a one-day symposium, where the investigators will present this report to the stakeholders including coordinators/managers decision-makers of health organizations and discuss implications and next steps for testing the platform more broadly across Canada and internationally with team's VITALISE network. In addition to traditional end-of-grant methods (e.g., conference presentations, open access publications), the investigators will also post regular updates and tailored executive summaries of findings on social media and on the CISSS and CIUSSS websites. This will be coupled with an end-of-project webinar to share results of the team's work. Training tools and sessions described above available online to help knowledge users build capacity for the use of the platform.

Data analysis Data will be analysed by type of stakeholder and program. The investigators will analyse the transcripts using content analysis techniques based on a deductive directed approach typically done in studies using the CFIR. While it will not be possible to sample for gender or sex in the composition of site implementation teams, the investigators will explore differences in the interview questions, analysis of qualitative data and modeling of quantitative data using participant self-identified gender. Sex and gender influence 1) behavior, 2) individual and organizational decision-making, 3) implementation and 4) may influence the platform design, how and why it is implemented, and use of the platform by clinicians and patient/families. As such the investigators will consider sex and gender in 1) development of knowledge tools for each site; 2) in development, usability testing, and interviews to evaluate facilitators and barriers and mechanisms for adoption and 3) in the usability testing in the design phase which will include 8 women and 8 men per stakeholder group (to explore gender/sex differences qualitatively).

Based on the one-year program indicators (2019-2020), the investigators have on average 569 patients with stroke and 393 with TBI, and total of 962 across the four regions and 8 programs. Data for all participants for the primary outcomes will be obtained from the SIPAD administrative database. It is anticipated a conservative estimate of 60% of patients (n=577) will consent and have complete data for research based on previous studies in the same settings and available to evaluate the secondary outcomes. In total, 28 managers and 60 clinicians across all programs were contacted. The investigators expect nearly 100% completion of questionnaires by clinicians as was found in a recent study in the programs.

Sample size:

The anticipated sample size is 8 programs (clusters) and a total of 962 participants for the primary outcome and 577 for the secondary outcomes. For the primary outcome, the study will have 80% power to detect standardized mean differences in direct rehabilitation time (primary outcome) of >=0.4 between control and implementation periods. This is based on a conservatively assumed intra-cluster correlation (ICC) of 0.20, and allowing for a coefficient of variation in cluster sizes of 0.42 (SD=50)/(mean=960/8=120),77,78 and taking the ICC and the design effect of 1.2 for cluster size variations ([1+(0.42^2+1)*120-1)*0.2] / [1+(120-1)*0.2] into consideration, the effective cluster size is n=100. This takes into account the stepped wedge design and the confounding effect of time (i.e. for a continuous outcome: time of direct rehabilitation; i.e. the investigators will be able to detect a change as small as 0.35 times the standard deviation of the outcome). The power calculations consider mixing both new patients and existing patients across trial steps (cluster autocorrelation=0.80). For the secondary outcomes, with a power of 90% the study will be able to detect a standardized effect size of >=0.50 (effective cluster size n=72/1.2 = 60 to account for heterogenous cluster sizes i.e. a total of 60 x 8 =480 observation points).

Apart from basic descriptive statistics, the analysis approach will be intention-to-treat using a generalize linear mixed effects (GLM) model. This model estimates the effect of order (intervention duration) on outcome accounting for clustered and correlated nature of the data (repeated assessments within nested levels of clusters: patients and sites which will be modeled as random effects). A log-link GLM will be employed to account for right-skewed time data (e.g. minutes per week and days of therapy). Estimated effects will be reported with 95% confidence intervals. For the secondary outcomes related to experience and health outcomes, a composite outcome approach will be used testing the effect of order on outcome independent of the source (experience) or measure (HRQL) used for that outcome. This approach increases power and reduces the need to consider multiple comparisons. As the effect of order (source, measure) may vary by time owing to secular effects, interaction terms with time will be included although not hypothesized to have a strong effect. Table 2 outlines the analysis plan for primary and secondary outcomes. The term for measures provides information on which measures are more contributing to the composite.

The general form of the model will be Outcome = order of randomization + time of assessment + order*time. The order*time interaction estimates whether the effect on the outcome of order (more or less exposure to the BRILLANT platform) depends on time which may happen if secular trends affect the impact of the intervention. Investigator's hypothesis is that this is unlikely, simplifying the analysis. For the secondary, experience outcomes and the HRQL outcomes, a composite analysis will be done where the source or measure is considered another cluster. The general form of the model is Outcome construct = Source (Who) [or Measure (What)] + Order + Time + Source [Measure]* Time which estimates whether time influences the association between the measure and outcome.

Economic evaluation will be performed only if an effect of intervention is detected. Additional data collection required is minimal as majority of cost data is from DPS database. Costs will be reported separately as: (1) provider time per patient, in hours by provider type; (2) healthcare utilization, measured as number of ED visits, number of hospitalizations, and hospital length of stay in days, obtained from DSP databases. Although services outside the organization may be missed, Quebec's regionalized healthcare mergers ensure that most patient services within a geographic area are captured. Although investigators may miss service utilization outside of the organization, because of mergers in Quebec, healthcare organizations include most services that one would use in a geographic area and as such, this approach should provide complete data.

Implementation analyses is needed to evaluate mechanisms for impact on outcome. Guided by Proctor's Framework the investigators will evaluate: relevance, acceptability by interview, meeting transcripts and the Technology Acceptance Measure (e.g. intention to use, perceived usefulness, and perceived ease of use), change in practice, feasibility, fidelity, and implementation cost (time for training, equipment); Platform Analytics and logs related to activity duration (comparing dates (first and last activities completed within each functionality), proportion (number of activities completed and total number of activities in each functionality), and clinical notes and communications on the platform will be analyzed thematically and presented descriptively.

Feasibility of implementing the platform There are three conditions in place that support successful implementation of the platform and trial feasibility. The first is stakeholder partnerships: the four health regions that will participate in this study are clinical partners of investigators' research center (CRIR), and each region has a lead investigator and knowledge user. The health regions acknowledges that they accept to be randomised to start using the platform in 2024/2025. The second is that many researchers have their research programs within the participant sites and are members of a larger digital health initiative, BRILLIANT (https://www.brilliant-cfi.ca/). Three of four health regions are a partner of the BRILLIANT CFI infrastructure (in-kind and cash contribution). The third condition, in parallel, there is a provincial mandate to implement Canadian ABI guidelines with local recommendations including standardized assessments and criteria for programs along the continuum of care. The researchers and clinicians participating in this study in each of the four health regions actively participated in the development and adaptation of recent ABI clinical guidelines adopted by the MSSS in 2015.

The guidelines are informing the reorganization of healthcare that will allow for continuity of care services, and more harmonized transitions at different levels of the healthcare system. Currently, the team is working with each region to implement clinical measures and patient reported outcome measures within the BRILLIANT Platform as part of the clinical workflow. The authors are implementing and evaluating the use of the MPAI measure to ensure that the impacts of ABI on physical, cognitive, emotional, behavioral, and social health are considered for rehabilitation planning.

Discussion This stepped wedge cluster randomized trial design aims to evaluate the impact of the BRILLIANT platform on intensity of rehabilitation, time to admission, health-related quality of life, and care experience for patients with cardiovascular and neurological conditions in Quebec's context. Without this trial, digital health platforms will be implemented in the health regions without evidence of their effectiveness. The scarcity of evidence on the mechanisms by which interventions work plagues implementation science. The investigators' longstanding clinical partnerships, the BRILLIANT infrastructure and the research network, provide an unprecedented opportunity for rehabilitation to: 1) inform decision-making in cardiovascular and neurological care by building in evidence-based guidelines in the reminders and recommendations to clinicians and patients; 2) provide evidence on if, and how digital health can improve cardiovascular and neurological best practices related to patient-centered care processes, assessment and treatment, and patient outcomes; 3) monitor the implementation process across health regions; 4) provide detailed mapping of the variability in the way the platform is implemented in each health region and across the cardiovascular and neurological care continuums (hospital, in- and outpatient rehabilitation) and serve as an exemplar to rehabilitation implementation teams; 5) if found to be effective, the trial will also measure the associated cost of implementation and cost savings (e.g., saved coordination and travel time) relative to the derived benefit from using the platform; 6) the implementation evaluation will provide information to inform the transferability and evaluation of the BRILLIANT platform internationally; and 7) when aggregated at a health region level, data from the BRILLIANT platform will inform quality improvement cycles, as part of a learning health system to identify processes and interventions that improve patient outcomes and health.

This study will provide valuable evidence on the effectiveness and feasibility of the BRILLIANT platform in improving rehabilitation care for patients with cardiovascular and neurological conditions. By addressing the challenges and pursuing future directions, the research team can contribute to improving patient outcomes and healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

Clinicians, coordinators, managers, working in the 8 participating programs.

Patients and caregivers must be able to:

* Provide informed consent to collect secondary outcomes (not needed for primary outcome, as identified administrative data will be provided by health regions)
* Speak and read English or French.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 962 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The intensity of rehabilitation | 27 months
  The intensity of rehabilitation (direct minutes of rehabilitation per week) will be calculated for all new patients seen during the control and intervention period using data from SIPAD64 (Système d'information pour les personnes ayant une déficience), that will be obtained from the directorate of professional services (DPS) administrative database where clinicians record the direct and indirect time spent with patients and caregivers.

SECONDARY OUTCOMES:
Time to be admitted to rehabilitation (inpatient or outpatient) | 12 months
  The time from cardiovascular or neurological condition onset to inpatient or home rehabilitation admission data will be obtained from SIPAD, similar to the primary outcome.
Health-related quality of life | 27 months
  Data from patients will be collected using the Quality of Life in Neurological Disorders (Neuro-QoL) battery of measures and the EuroQol 5-Dimension, 5-Level (EQ-5D-5L). The EQ-5D-5L index score ranges from -0.281 to 1.000, with higher scores indicating "full health-related quality of life". The Neuro-QoL instruments each yield standardized T-scores ranging from 10 to 90 (mean 50, SD 10 in the reference population), where higher scores indicate more of the concept being measured. Caregivers' health-related quality of life will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS-29) Profile, which produces domain scores standardized to a T-score metric (mean 50), ranging from 20 to 80. Higher scores reflect more of the domain, with better outcomes for positive domains and worse outcomes for negative domains.
Care experience, and perceived effectiveness | 27 months
  Caregiver burden will be measured with the Bakas Caregiving Outcomes Scale (15 items, scores 15 - 105; in which higher scores represent more negative change in well-being). Patient experience will be assessed using the Patient Participation in Rehabilitation Questionnaire (scores 0 - 100; in which higher scores represent greater participation). Clinicians' experience implementing BRILLIANT will be measured using the Normalization Measure Development (NoMAD, scores 20 - 100; in which higher scores represent greater normalization of practice change).
Sex and gender identification | 27 months
  Sex and gender identification will be collected using two self-identified items.
Satisfaction with the BRILLIANT Platform | 12 months
  Satisfaction with the BRILLIANT Platform will be explored in semi-structured interviews with 20 clinicians, 4 managers, and 40 patients/caregivers, focusing on usability and improvements.
Economic evaluation - cost-utility analysis | 27 months
  For cost-utility analysis, Quality-Adjusted Life Years (QALYs) will be estimated from the EQ-5D-5L (index scores range -0.281 to 1.000).
Economic evaluation - cost-effectiveness | 27 months
  Incremental cost-effectiveness ratios (ICERs) will be calculated from the Ministry of Health and Social Services perspective.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CIUSSS du Centre-Sud-de-l'Île-de-Montréal, Montreal, Quebec
  - Centre de réadaptation Lethbridge-Layton-Mackay, installation Constance-Lethbridge, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmed S, Archambault P, Auger C, Durand A, Fung J, Kehayia E, Lamontagne A, Majnemer A, Nadeau S, Pineau J, Ptito A, Swaine B. Biomedical Research and Informatics Living Laboratory for Innovative Advances of New Technologies in Community Mobility Rehabilitation: Protocol for Evaluation and Rehabilitation of Mobility Across Continuums of Care. JMIR Res Protoc. 2022 Jun 1;11(6):e12506. doi: 10.2196/12506. PMID 35648455
- [Background] 2. Canadian stroke for best practices "Csbp". Recommendations: Overview, Methods and Knowledge Exchange. https://www.strokebestpractices.ca/recommendations
- [Background] 3. Institut national d'excellence en santé et en services sociaux- Ontario neurotrauma foundation "INESSS-ONF". Clinical practice for the rehabilitation of adults with moderate to severe TBI. https://braininjuryguidelines.org/modtosevere/
- [Background] 4. Statistics Canada. Table 102-0561 - Leading causes of death, total population, by age group and sex, Canada. CANSIM (death database) [Internet]. Ottawa (Ontario): Statistics Canada. 2017;
- [Background] 5. Ministère de la Santé et des Sevices sociaux (MSSS). Continuum de services pour les personnes à risque de subir ou ayant subi un accident vasculaire cérébral: Plan de mise en œuvre Phase 2016-2018. 2016: Québec. p. 1-64.
- [Background] Langhorne P, Collier JM, Bate PJ, Thuy MN, Bernhardt J. Very early versus delayed mobilisation after stroke. Cochrane Database Syst Rev. 2018 Oct 16;10(10):CD006187. doi: 10.1002/14651858.CD006187.pub3. PMID 30321906
- [Background] 7. Publications du ministère de la Santé et des Services sociaux "MSSS". Trousse d'outils cliniques pour l'évaluation des personnes ayant subi un accident vasculaire cérébral (AVC) - Phases hyperaiguë et aiguë de l'AVC. https://publications.msss.gouv.qc.ca/msss/document-002419/?&txt=personne&msss_valpub&date=DESC
- [Background] 8. Publications du ministère de la Santé et des Services sociaux "MSSS". Continuum de services pour les personnes à risque de subir ou ayant subi un accident vasculaire cérébral Paramètres organisationnels de réadaptation, réintégration et de maintien dans la communauté en AVC. 2021. https://publications.msss.gouv.qc.ca/msss/fichiers/2017/17-944-02W.pdf
- [Background] Alhasani R, Auger C, Paiva Azevedo M, Ahmed S. Quality of mobility measures among individuals with acquired brain injury: an umbrella review. Qual Life Res. 2022 Sep;31(9):2567-2599. doi: 10.1007/s11136-022-03103-4. Epub 2022 Mar 11. PMID 35275377
- [Background] Alhasani R, Godbout M, Durand A, Auger C, Lamontagne A, Ahmed S. Informing the development of an outcome set and banks of items to measure mobility among individuals with acquired brain injury using natural language processing. BMC Neurol. 2022 Dec 9;22(1):464. doi: 10.1186/s12883-022-02938-1. PMID 36494770
- [Background] Alhasani R, Radman D, Auger C, Lamontagne A, Ahmed S. Clinicians and individuals with acquired brain injury perspectives about factors that influence mobility: creating a core set of mobility domains among individuals with acquired brain injury. Ann Med. 2021 Dec;53(1):2365-2379. doi: 10.1080/07853890.2021.2015539. PMID 34894914
- [Background] 12. Alhasani R, Radman, D., Auger, C., Lamontagne, A., Ahmed, S. . Clinicians', Patients' and Caregivers' Perspectives about Service Provision across the Continuum of Care to Improve Mobility and Participation among Individuals with Acquired Brain Injury. . Submitted to Qualitative Health Research Journal. Submitted February 11, 2021
- [Background] 13. Alhasani R, Ferreira, T. J., Valois, M-F., Alghamdi, S. Singh, D. Ahmed, S. . Enrollment and dropout rates of individuals with chronic obstructive pulmonary disease approached in telehealth interventions: A systematic review and meta-analysis. Submitted to Chest Journal Submitted on March 8, 2021
- [Background] Lam Wai Shun P, Swaine B, Bottari C. Clinical reasoning underlying acute care occupational therapists' assessment of rehabilitation potential after stroke or brain injury: A constructivist grounded theory study. Aust Occup Ther J. 2022 Apr;69(2):177-189. doi: 10.1111/1440-1630.12781. Epub 2021 Dec 22. PMID 34939206
- [Background] Borgen IMH, Roe C, Brunborg C, Tenovuo O, Azouvi P, Dawes H, Majdan M, Ranta J, Rusnak M, Wiegers EJA, Tverdal C, Jacob L, Cogne M, von Steinbuechel N, Andelic N; CENTER-TBI participants investigators. Care transitions in the first 6months following traumatic brain injury: Lessons from the CENTER-TBI study. Ann Phys Rehabil Med. 2021 Nov;64(6):101458. doi: 10.1016/j.rehab.2020.10.009. Epub 2021 Jul 23. PMID 33246186
- [Background] Fann JR, Hart T, Ciol MA, Moore M, Bogner J, Corrigan JD, Dams-O'Connor K, Driver S, Dubiel R, Hammond FM, Kajankova M, Watanabe TK, Hoffman JM. Improving transition from inpatient rehabilitation following traumatic brain injury: Protocol for the BRITE pragmatic comparative effectiveness trial. Contemp Clin Trials. 2021 May;104:106332. doi: 10.1016/j.cct.2021.106332. Epub 2021 Feb 27. PMID 33652127
- [Background] McNair ND. The Projected Transition Trajectory for Survivors and Carers of Patients Who Have Had a Stroke. Nurs Clin North Am. 2019 Sep;54(3):399-408. doi: 10.1016/j.cnur.2019.04.008. Epub 2019 Jun 8. PMID 31331626
- [Background] Moore JL, Nordvik JE, Erichsen A, Rosseland I, Bo E, Hornby TG; FIRST-Oslo Team. Implementation of High-Intensity Stepping Training During Inpatient Stroke Rehabilitation Improves Functional Outcomes. Stroke. 2020 Feb;51(2):563-570. doi: 10.1161/STROKEAHA.119.027450. Epub 2019 Dec 30. PMID 31884902
- [Background] Hebert D, Lindsay MP, McIntyre A, Kirton A, Rumney PG, Bagg S, Bayley M, Dowlatshahi D, Dukelow S, Garnhum M, Glasser E, Halabi ML, Kang E, MacKay-Lyons M, Martino R, Rochette A, Rowe S, Salbach N, Semenko B, Stack B, Swinton L, Weber V, Mayer M, Verrilli S, DeVeber G, Andersen J, Barlow K, Cassidy C, Dilenge ME, Fehlings D, Hung R, Iruthayarajah J, Lenz L, Majnemer A, Purtzki J, Rafay M, Sonnenberg LK, Townley A, Janzen S, Foley N, Teasell R. Canadian stroke best practice recommendations: Stroke rehabilitation practice guidelines, update 2015. Int J Stroke. 2016 Jun;11(4):459-84. doi: 10.1177/1747493016643553. Epub 2016 Apr 14. PMID 27079654
- [Background] 20. Simmons-Mackie N, Worrall L, Murray LL, et al. The top ten: best practice recommendations for aphasia. Aphasiology. 2017;31(2):131-151.
- [Background] Ross SY, Roberts S, Taggart H, Patronas C. Stroke Transitions of Care. Medsurg Nurs. 2017 Mar;26(2):119-23. PMID 30304593
- [Background] Oyesanya TO, Loflin C, Harris G, Bettger JP. "Just tell me in a simple way": A qualitative study on opportunities to improve the transition from acute hospital care to home from the perspectives of patients with traumatic brain injury, families, and providers. Clin Rehabil. 2021 Jul;35(7):1056-1072. doi: 10.1177/0269215520988679. Epub 2021 Jan 20. PMID 33472414
- [Background] Tighe SA, Ball K, Kensing F, Kayser L, Rawstorn JC, Maddison R. Toward a Digital Platform for the Self-Management of Noncommunicable Disease: Systematic Review of Platform-Like Interventions. J Med Internet Res. 2020 Oct 28;22(10):e16774. doi: 10.2196/16774. PMID 33112239
- [Background] Liddy C, Keely E. Using the Quadruple Aim Framework to Measure Impact of Heath Technology Implementation: A Case Study of eConsult. J Am Board Fam Med. 2018 May-Jun;31(3):445-455. doi: 10.3122/jabfm.2018.03.170397. PMID 29743227
- [Background] Bodenheimer T, Sinsky C. From triple to quadruple aim: care of the patient requires care of the provider. Ann Fam Med. 2014 Nov-Dec;12(6):573-6. doi: 10.1370/afm.1713. PMID 25384822
- [Background] Hemming K, Taljaard M. Reflection on modern methods: when is a stepped-wedge cluster randomized trial a good study design choice? Int J Epidemiol. 2020 Jun 1;49(3):1043-1052. doi: 10.1093/ije/dyaa077. PMID 32386407
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] 30. Ku B, Lupton E. Health Design Thinking: Creating Products and Services for Better Health. MIT Press; 2020.
- [Background] Roberts JP, Fisher TR, Trowbridge MJ, Bent C. A design thinking framework for healthcare management and innovation. Healthc (Amst). 2016 Mar;4(1):11-4. doi: 10.1016/j.hjdsi.2015.12.002. Epub 2016 Jan 14. PMID 27001093
- [Background] 32. Vaisman A. An introduction to business process modeling. Springer; 2012:29-61.
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Varsi C, Ekstedt M, Gammon D, Ruland CM. Using the Consolidated Framework for Implementation Research to Identify Barriers and Facilitators for the Implementation of an Internet-Based Patient-Provider Communication Service in Five Settings: A Qualitative Study. J Med Internet Res. 2015 Nov 18;17(11):e262. doi: 10.2196/jmir.5091. PMID 26582138
- [Background] Kengne Talla P, Thomas A, Ataman R, Auger C, McKerral M, Wittich W, Poncet F, Ahmed S. Evaluating the implementation of the Mayo-Portland Adaptability Inventory-4 (MPAI-4) in three rehabilitation settings in Quebec: a mixed-methods study protocol. BMJ Open. 2023 May 23;13(5):e068866. doi: 10.1136/bmjopen-2022-068866. PMID 37221032
- [Background] Perry CK, Damschroder LJ, Hemler JR, Woodson TT, Ono SS, Cohen DJ. Specifying and comparing implementation strategies across seven large implementation interventions: a practical application of theory. Implement Sci. 2019 Mar 21;14(1):32. doi: 10.1186/s13012-019-0876-4. PMID 30898133
- [Background] (MSSS) MdlSedSs. SIPAD - Système d'information pour les personnes ayant une déficience. 2021. http://www.ti.msss.gouv.qc.ca/getdoc/8fce570f-c353-4a39-b332-bee5ca1b9eec/SIPAD.aspx
- [Background] 39. Ministère de la Santé et des Sevices sociaux (MSSS). L'implantation d'un système de suivi global et intégré de la performance du programme-services Déficience physique. 2016;
- [Background] 40. Vanderbilt Redcap.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Cella D, Lai JS, Nowinski CJ, Victorson D, Peterman A, Miller D, Bethoux F, Heinemann A, Rubin S, Cavazos JE, Reder AT, Sufit R, Simuni T, Holmes GL, Siderowf A, Wojna V, Bode R, McKinney N, Podrabsky T, Wortman K, Choi S, Gershon R, Rothrock N, Moy C. Neuro-QOL: brief measures of health-related quality of life for clinical research in neurology. Neurology. 2012 Jun 5;78(23):1860-7. doi: 10.1212/WNL.0b013e318258f744. Epub 2012 May 9. PMID 22573626
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Sikorskii A, Victorson D, O'Connor P, Hankin V, Safikhani A, Crane T, Badger T, Wyatt G. PROMIS and legacy measures compared in a supportive care intervention for breast cancer patients and caregivers: Experience from a randomized trial. Psychooncology. 2018 Sep;27(9):2265-2273. doi: 10.1002/pon.4825. Epub 2018 Jul 17. PMID 29956396
- [Background] Bakas T, Champion V. Development and psychometric testing of the Bakas Caregiving Outcomes Scale. Nurs Res. 1999 Sep-Oct;48(5):250-9. doi: 10.1097/00006199-199909000-00005. PMID 10494909
- [Background] 46. Badgett ML, Baker K, Conron K, et al. Best practices for asking questions to identify transgender and other gender minority respondents on population-based surveys (GenIUSS). The GenIUSS Group, UCLA Williams Institute. 2014;
- [Background] Lindberg J, Kreuter M, Person LO, Taft C. Patient Participation in Rehabilitation Questionnaire (PPRQ)-development and psychometric evaluation. Spinal Cord. 2013 Nov;51(11):838-42. doi: 10.1038/sc.2013.98. Epub 2013 Sep 17. PMID 24042990
- [Background] 48. Finch T, Girling M, May C, et al. NoMAD: implementation measure based on Normalization Process Theory.[Measurement instrument]. 2015.
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] 50. Pilote L. GENESIS-PRAXY Questionnaire. https://cihr-irsc.gc.ca/e/50529.html
- [Background] Kontos E, Blake KD, Chou WY, Prestin A. Predictors of eHealth usage: insights on the digital divide from the Health Information National Trends Survey 2012. J Med Internet Res. 2014 Jul 16;16(7):e172. doi: 10.2196/jmir.3117. PMID 25048379
- [Background] Auger C, Miller WC, Jutai JW, Tamblyn R. Development and feasibility of an automated call monitoring intervention for older wheelchair users: the MOvIT project. BMC Health Serv Res. 2015 Sep 16;15:386. doi: 10.1186/s12913-015-1048-0. PMID 26376853
- [Background] 53. Ahmed S PT, D Kairy, A Rochette. Use of telehealth during COVID in an Early Assisted Discharge Program Post-Stroke. Submitted PlOS One. February 2022.;
- [Background] Voldal EC, Hakhu NR, Xia F, Heagerty PJ, Hughes JP. swCRTdesign: An RPackage for Stepped Wedge Trial Design and Analysis. Comput Methods Programs Biomed. 2020 Nov;196:105514. doi: 10.1016/j.cmpb.2020.105514. Epub 2020 May 21. PMID 32554025
- [Background] 55. Stepped Wedge Power Calculation, Shiny app 2021. https://swcrtdesign.shinyapps.io/stepped_wedge_power_calculation/
- [Background] 56. Hemming K, Girling A, Haines T, Lilford R. Protocol: Consort extension to stepped wedge cluster randomised controlled trial. BMJ. 2014;
- [Background] Hemming K, Kasza J, Hooper R, Forbes A, Taljaard M. A tutorial on sample size calculation for multiple-period cluster randomized parallel, cross-over and stepped-wedge trials using the Shiny CRT Calculator. Int J Epidemiol. 2020 Jun 1;49(3):979-995. doi: 10.1093/ije/dyz237. PMID 32087011
- [Background] McCoy CE. Understanding the Use of Composite Endpoints in Clinical Trials. West J Emerg Med. 2018 Jul;19(4):631-634. doi: 10.5811/westjem.2018.4.38383. Epub 2018 Jun 4. PMID 30013696
- [Background] Pogue J, Devereaux PJ, Thabane L, Yusuf S. Designing and analyzing clinical trials with composite outcomes: consideration of possible treatment differences between the individual outcomes. PLoS One. 2012;7(4):e34785. doi: 10.1371/journal.pone.0034785. Epub 2012 Apr 17. PMID 22529934
- [Background] Geng EH, Baumann AA, Powell BJ. Mechanism mapping to advance research on implementation strategies. PLoS Med. 2022 Feb 8;19(2):e1003918. doi: 10.1371/journal.pmed.1003918. eCollection 2022 Feb. PMID 35134069
- [Background] Holden RJ, Karsh BT. The technology acceptance model: its past and its future in health care. J Biomed Inform. 2010 Feb;43(1):159-72. doi: 10.1016/j.jbi.2009.07.002. Epub 2009 Jul 15. PMID 19615467
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Teasell R, Salbach NM, Foley N, Mountain A, Cameron JI, Jong A, Acerra NE, Bastasi D, Carter SL, Fung J, Halabi ML, Iruthayarajah J, Harris J, Kim E, Noland A, Pooyania S, Rochette A, Stack BD, Symcox E, Timpson D, Varghese S, Verrilli S, Gubitz G, Casaubon LK, Dowlatshahi D, Lindsay MP. Canadian Stroke Best Practice Recommendations: Rehabilitation, Recovery, and Community Participation following Stroke. Part One: Rehabilitation and Recovery Following Stroke; 6th Edition Update 2019. Int J Stroke. 2020 Oct;15(7):763-788. doi: 10.1177/1747493019897843. Epub 2020 Jan 27. PMID 31983296
- [Background] Mountain A, Patrice Lindsay M, Teasell R, Salbach NM, de Jong A, Foley N, Bhogal S, Bains N, Bowes R, Cheung D, Corriveau H, Joseph L, Lesko D, Millar A, Parappilly B, Pikula A, Scarfone D, Rochette A, Taylor T, Vallentin T, Dowlatshahi D, Gubitz G, Casaubon LK, Cameron JI. Canadian Stroke Best Practice Recommendations: Rehabilitation, Recovery, and Community Participation following Stroke. Part Two: Transitions and Community Participation Following Stroke. Int J Stroke. 2020 Oct;15(7):789-806. doi: 10.1177/1747493019897847. Epub 2020 Jan 27. PMID 31983292
- [Background] 66. Malec J. The Mayo Portland Adaptability Inventory: The Center for Outcome Measurement in Brain Injury; 2005. 2014.
- [Background] Ministère de la Santé et des Sevices sociaux (MSSS). Continuum de services pour les personnes à risque de subir ou ayant subi un accident vasculaire cérébral 2018: Quebec. p. 1-89.
- [Background] Sicotte C, Pare G. Success in health information exchange projects: solving the implementation puzzle. Soc Sci Med. 2010 Apr;70(8):1159-65. doi: 10.1016/j.socscimed.2009.11.041. Epub 2010 Feb 4. PMID 20137847